CLINICAL TRIAL: NCT03469505
Title: Cooperative Pain Education and Self-management: Expanding Treatment for Real-world Access (COPES ExTRA)
Acronym: COPES ExTRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000024225; 1UG3AT009767-01 (NIH); 4UH3AT009767-03 (NIH)
Record Dates: First submitted 2018-02-02; First posted 2018-03-19 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Pain, Chronic
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- data from veterans using COPES (Active Comparator): Data from veterans using COPES for chronic pain
  Interventions: Behavioral: COPES
- data from veterans using CBT-CP (Active Comparator): Data from veterans using CBT-CP for chronic pain
  Interventions: Behavioral: CBT-CP

INTERVENTIONS:
Behavioral: COPES — Cooperative Pain Education and Self-Management for chronic pain therapy.
  Arms: data from veterans using COPES
Behavioral: CBT-CP — Cognitive Behavioral Therapy for Chronic Pain
  Arms: data from veterans using CBT-CP

SUMMARY:
To conduct a superiority trial of COPES versus standard Veterans Health Administration (VHA) Cognitive Behavioral Therapy Chronic Pain (CBT-CP)

DETAILED DESCRIPTION:
Our prior efficacy trial found that COPES was not inferior to in-person CBT-CP and that participants attended, on average, a little over two more treatment weeks in COPES than in-person treatment, presumably due to the ease of in-home treatment attendance relative to in-person treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic musculoskeletal pain receiving care in VHA.
* A pain-related musculoskeletal diagnosis indicated by an EHR identified ICD-9 or -10 code.
* The presence of chronic pain of at least moderate severity with EHR NRS pain scores ≥ 4 in three separate months for a period of 12 months.
* Absence of mental illness serious enough to have resulted in an inpatient psychiatric hospitalization in the prior 3 months excluding detoxification of alcohol or drugs.
* Absence of malignant cancer diagnosis or receipt of hospice or end-of-life palliative care.
* Ability to participate safely in the walking portion of the intervention as evidenced by patient-reported ability to walk at least one block and absence of diabetic foot ulcers at the time of the enrollment.
* Absence of significant cognitive impairment as identified by a dementia-related diagnosis.
* Availability of a touch-tone land-line or cellular telephone and no vision or hearing deficits that would impair participation verified by patient report at the time of the enrollment call.

Exclusion Criteria:

* Patients not fitting criteria for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 764 (Actual)
Dates: Start 2019-12-27 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Brief Pain Inventory, Interference Subscale Score | 4 months
  The Brief Pain Inventory Interference Score is patient-reported pain-related interference. Data will be collected through automated IVR calls.

SECONDARY OUTCOMES:
The Brief Pain Inventory, Interference Score | 6 months, 12 months
  The Brief Pain Inventory Interference Score is patient-reported pain-related interference. Data will be collected through automated IVR calls.
Numeric Rating Score, Pain Intensity | 4 month
  The single average pain intensity rating question from the self-reported, Brief Pain Inventory. Data will be collected through automated IVR calls.
PEG-3 | 4 month
  A Three-Item Scale Assessing Pain Intensity and Interference. Data will be collected through automated IVR calls.
Depression symptom severity | 4 months
  Depression symptom severity will be assessed using the 8-item Patient Health Questionnaire (PHQ-8) a widely-used measure with excellent internal consistency and stability. Data will be collected through an automated IVR.
Pain Catastrophizing Scale- Short Form | 4 months
  The Pain Catastrophizing Scale (PCS)-Short Form is a validated, 3-item self-report scale that examines thoughts and feelings people may experience when they are in pain. Data will be collected through an automated IVR
Sleep Quality | 4 months
  Sleep quality will be measured using the Insomnia Severity Index and will assess subjective sleep quality. Data will be collected through automated IVR calls.
Pain Self-Efficacy | 4 months
  Self-Efficacy will be assessed using 1-Item of the Pain Self-Efficacy Questionnaire. Data will be collected through automated IVR calls.
Patient Global Perception of Change | 4 months
  The Patient Global Perception of Change scale is a single item measure that quantifies a participant's overall perception of improvement since beginning treatment and the clinical importance of that improvement. Participants indicate improvement on a 7 point "much worse" to "much better" scale. Data will be collected through automated IVR calls.
Pain Satisfaction Questionnaire | 4 month
  Pain satisfaction will be measured using an adapted Pain Satisfaction Questionnaire. This 5-item measure about patient self report of experience of treatment . Data will be collected through automated IVR calls.
Treatment dose | Up to 12 months post baseline
  Number of cognitive behavioral therapy for chronic pain sessions attended for this treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Heapy, Phd, Principal Investigator — VA Office of Research and Development
Locations (9):
- United States (9):
  - Edward Hines, Jr. VA Hospital, Hines, Illinois
  - VA Central Western Massachusetts, Leeds, Massachusetts
  - VA Ann Arbor Healthcare System, Ann Arbor, Michigan
  - G.V. (Sonny) Montgomery VA Medical Center, Jackson, Mississippi
  - Oklahoma City VA Health Care System, Oklahoma City, Oklahoma
  - Ralph H. Johnson VA Medical Center, Charleston, South Carolina
  - VA North Texas Healthcare System, Dallas, Texas
  - VA Central Texas Healthcare System, Temple, Texas
  - VA Puget Sound Healthcare System, Seattle, Washington